CLINICAL TRIAL: NCT03492892
Title: Use of Metabolomics to Differentiate the Antihypertensive Effect of Acupuncture From Sham Acupuncture in Hypertensives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012KL-003
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Hypertension,Essential
Keywords: acupuncture; hypertension; targeted metabolome; pilot clinical trial
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Use real acupuncture treatment for blood pressure management in patients with hypertension
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): Use non-acupoint as the stimulating site in acupuncture for the treatment of hypertension
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — Stimulate acupoint with filiform needles to restore the healthy condition of patients
  Arms: Acupuncture
Device: Sham Acupuncture — Stimulate non-acupoint with filiform needles to treat the condition of patients
  Arms: Sham Acupuncture

SUMMARY:
To assess the effect of acupuncture versus sham acupuncture on regulating the targeted metabolome of hypertensive patients.

DETAILED DESCRIPTION:
Acupuncture has been widely used for blood pressure management. Its effect on the cardiovascular-related targeted metabolome is still unknown. This pilot study aimed to assess the effect of acupuncture versus sham acupuncture on regulating the targeted metabolome of hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* aged between 45 and 75 years;
* were diagnosed as stage I hypertension in the first visit, or used to be diagnosed with stage I hypertension in recent 1 year, but without any medication history;
* without neurological, other cardiovascular, hepatic and renal disease, and other visceral diseases;
* the basal metabolism rate of a patient, which was measured by the retrospective dietary questionnaire at baseline, should be approximately 1:1.4;
* didn't administer any drugs or herbs in at 15 days before the start of the study;
* didn't participate in any study other than this;
* agreed to cooperate with researchers in all research procedures after they were introduced this study; and
* provided with written informed consent.

Exclusion Criteria:

* age≤45 or age≥75;
* with hypertension which was secondary to other diseases, such as renal vascular disease, Cushing's syndrome, hyperadrenocorticism and drug-induced hypertension;
* had complicated cardiovascular, digestive, respiratory, urinary, blood, nervous, endocrine system and other severe primary diseases and failed to effectively control in clinic;
* accompanied by epilepsy, sleep apnea, hypopnea syndrome, etc.;
* with psychiatric symptoms such as severe depression or anxiety (SAS≥70, or SDS≥72);
* pregnant or lactating woman, or woman of reproductive age who was intended to conceive in recent 1 year;
* with abnormality in laboratory test of blood biochemistry, or with contagious risks, such as HIV virus carrier, or patient with positive Hepatitis B Virus (HBV) superficial antigen;
* with malignant tumor or other severe consuming diseases, or patients with infections or bleeding disorders;
* alcoholics or drug abusers, or vegetarians;
* used to suffer from acute diseases in recent 2 weeks, such as high fever, or gastritis;
* used to administer any drug that may potentially impaired renal or hepatic function;
* with cardiovascular disease that had been treated with acupuncture within recent three months; or
* undergoing other clinical trials.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-08-19 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
24 hour ambulatory blood pressure | up to week 6

SECONDARY OUTCOMES:
targeted plasma metabolome | up to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Fan-rong Liang, Prof., Principal Investigator — Chengdu University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data will be shared upon request.